CLINICAL TRIAL: NCT04020107
Title: Validity of Somatosensori Remediation for Postural Control in the Treatment of Ehlers-Danlos Syndrome Hypermobility Type (hEDS)
Acronym: VITALISED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-2012
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Ehlers-Danlos Syndrome Hypermobility Type (hEDS)
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compressive garment associated with physical therapy (Active Comparator)
  Interventions: Other: Compressive garment and Somatosensori Remediation
- Low compressive garment associated with physical therapy (Placebo Comparator)
  Interventions: Other: Compressive garment and Somatosensori Remediation

INTERVENTIONS:
Other: Compressive garment and Somatosensori Remediation — Each patient will benefit successively: from a classic care, over a period of 2 to 4 months, then will be treated with compressive or low compressive garments associated with specific proprioceptive physiotherapy program during the next 4 months. Finally, the 4 last months, patient will made adapted physical activity with both dance sessions strengthening the body diagram and stretching sessions

SUMMARY:
In the absence of a medical consensus, the current management of Ehlers-Danlos Syndrome hypermobility type (hEDS) remains very speculative That's why investigators want in this study to demonstrate the beneficial contribution of an innovative therapeutic strategy combining reprogramming and substitution somatosensory. This therapy is based primarily on the somesthetic substitution provided by compression garments(VC). Indeed, the VC port associated with stimulation of the somesthetic system via a specific program of physiotherapy (e.e. centered on body awareness through movement) could potentiate the effectiveness of care, and therefore enhance its long-term beneficial effect. The patient could thus regain his mobility, his functional independence, and thus considerably increase its quality of life. Thereafter, the practice of an adapted physical activity (APA), by the sensory stimulation induced and its playful nature, will allow patients to preserve and sustain the benefits of taking load previously carried out. Validation of this therapeutic approach would offer an effective solution may subsequently be proposed to the entire medical profession as reference support in the treatment of the hEDS.

This study plans to include, over a period of two years, 40 patients with hypermobile Ehlers-Danlos syndrome and 40 healthy volunteers controls. Patients will be followed for a period of one year divided into 3 periods of 4 months, between which they will be evaluated in order to quantify the impact of the intervention performed at each stage of the protocol.

Each patient will benefit successively: from a classic care, over a period of 2 to 4 months, then will be treated with compressive garments or with low compressive garment during the next 4 months in association with proprioceptive physical therapy. Finally, the 4 last months, patient will participate in an APA with both dance sessions strengthening the body diagram and stretching sessions.

The aim of this work is therefore to evaluate the effect of a treatment specifically oriented towards somatosensory remediation.

ELIGIBILITY:
Inclusion Criteria:

For EDS patients :

* Subjects aged 18 to 40,
* SEDh patients newly diagnosed for less than 2 years according to international criteria of 2017,
* Having a Body Mass Index (BMI) of less than 30,
* Affiliated to a social security scheme,
* Having read the information document and given in writing their free and informed consent to participate in the study.

For healthy volunteers :

* Subjects aged 18 to 40,
* Having a Body Mass Index (BMI) of less than 30,
* Having a Beigthon score <5 (no joint hypermobility),
* Having normal muscle strength,
* Affiliated to a social security scheme,
* Having read the information document and given in writing their free and informed consent to participate in the study.

Exclusion Criteria:

For EDS patients :

* Subjects under 18,
* Proprioceptive physiotherapy (Huber 360 platform type, LPG) in progress or already performed,
* previous treatment of hEDS capable of limiting the effects of rehabilitation (e.g. orthodontics, orthoptics),
* Diagnosis of other connective tissue abnormalities,
* Earlier prescription of compression garments,
* Pregnant or lactating women,
* Lack of effective contraception during the study period for women
* Person under tutorship or curatorship, or deprived of liberty by judicial or administrative decision,
* Mental or physical impossibility to agree to participate in the study,
* Known allergy to one of the components of compression garments,
* Disabling motor impairment, or limiting the performance of motor and psychomotor tests.
* Simultaneous participation in another clinical study.

For healthy volunteers :

* Subjects under 18,
* History of vascular, neurological, musculoskeletal or vestibular disorders,
* Having orthoptic, orthopedic or orthodontic disorders,
* Previous history or progressive disease of vascular, ophthalmological, neurological, musculoskeletal condition, or vestibular condition
* Pregnant or lactating women,
* Person under tutorship or curatorship, or deprived of liberty by judicial or administrative decision,
* Mental or physical impossibility to agree to participate in the study,
* Simultaneous participation in another clinical study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
analysis of center of pressure displacements on force platform | at month 8
  The main evaluation criterion is the complexity of postural control after 8 months of treatment (M8) through an analysis of the organization postural fluctuations (i.e. analysis of center of pressure displacements on force platforms6).

CONTACTS AND LOCATIONS:
Locations (1):
- Caen Univerity Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No